CLINICAL TRIAL: NCT04661449
Title: Childhood Health Outcomes in Term, Large-for-gestational-age Infants: Effects of Lifestyle Intervention in the Postnatal First Year
Brief Title: Effects of Lifestyle Intervention on Childhood Outcomes in LGA Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: XH-20-023
Record Dates: First submitted 2020-11-01; First posted 2020-12-10 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2020-12

CONDITIONS: Childhood Overweight
Keywords: large for gestational age
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Intervention (Experimental): every 3 months within 1 year.
  Interventions: Other: Comprehensive lifestyle intervention
- control group (No Intervention): Regular follow-up every 6 months within 1 year.

INTERVENTIONS:
Other: Comprehensive lifestyle intervention — Feeding guidance: promoting exclusive breastfeeding and healthy diet (Pediatrician). Motor development assessment and guidance: Alberta Infant movement scale (AIMS) evaluation, guidance for motor development (Rehabilitation Therapist). Healthcare education: improvement of environmental exposure (Pediatrician).
  Arms: Lifestyle Intervention

SUMMARY:
Large-for-gestational-age (LGA) infants have a higher risk of metabolic disease later in life, and their postnatal growth in early childhood may be associated with long-term adverse outcomes. The purpose of this study is to explore whether comprehensive lifestyle intervention in the first year after birth in LGA infants will reduce the rate of overweight/obesity at childhood and improve neurodevelopmental outcomes and its possible mechanism.

DETAILED DESCRIPTION:
Term LGA infants will be randomly divided into two groups shortly after birth: intervention group and control group. Infants in intervention group will attend the follow-up clinic and motor development assessment and guidance will be provided every three months in the first year. Other lifestyle interventions include feeding guidance and healthcare education. Infants in control group will routinely attend the follow-up clinic every six months. Primary outcome is the rate of overweight/obesity at two years old and seven years old. Neurodevelopmental assessment, carotid intima-media thickness (CIMT) and blood pressure at childhood will also be evaluated. The association of the outcome of LGA infants at two years old and the biomarkers in cord blood will be investigated, which includes serum leptin, insulin, insulin-like growth factors -1 (IGF-1), blood lipid series and adiponectin.

ELIGIBILITY:
Inclusion Criteria:

* term
* large-for-gestational-age infants

Exclusion Criteria:

* major genetic disorder
* congenital anomalies
* severe digestive disease

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 138 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Rate of overweight/obesity at 2 years old | at 2 years old
  Weight and height will be combined to report BMI in kg/m^2. According to the intergrowth-21st age-specific BMI standard issued in 2014, BMI ≥ 85th percentile is defined as overweight; BMI ≥ 95th percentile is defined as obesity
Rate of overweight/obesity at 7 years old | at 7 years old
  Weight and height will be combined to report BMI in kg/m^2. According to the intergrowth-21st age-specific BMI standard issued in 2014, BMI ≥ 85th percentile is defined as overweight; BMI ≥ 95th percentile is defined as obesity

SECONDARY OUTCOMES:
Neurodevelopmental assessment at 2 years old | at 2 years old
  Bayley III's assessment of infants is divided into five areas: cognition, language, body movement, social emotion and adaptive behavior.
Carotid intima-media thickness (CIMT) at 2 years old | at 2 years old
  Carotid intima-media thickness (CIMT) will be measured by experienced Pediatric Cardiologist.
Association of BMI at 2 years old with biomarkers in cord blood | at 2 years old
  Biomarkers include: serum leptin, insulin, IGF - Ⅰ, blood lipid series, adiponectin
Association of BMI at 7 years old with biomarkers in cord blood | at 7 years old
  Biomarkers include: serum leptin, insulin, IGF - Ⅰ, blood lipid series, adiponectin
Blood pressure at 7 years old | at 7 years old
  Blood pressure will be measured by experienced nurses.
Carotid intima-media thickness (CIMT) at 7 years old | at 7 years old
  Carotid intima-media thickness (CIMT) will be measured by experienced Pediatric Cardiologist.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital, Shanghai, Shanghai Municipality, China